CLINICAL TRIAL: NCT04740125
Title: PSYCHOLOGICAL IMPACT, STRESS FACTORS AND BEHAVIOURS IN HEALTH CARE PROFESSIONALS DURING THE COVID-19 PANDEMIC IN TUNISIA
Brief Title: SURVEY ABOUT STRESS-COVID IN HEALTH CARE WORKERS IN NORTH AFRICA COUNTRY
Acronym: COVID-STRESS
Status: Completed | Type: Observational
Sponsor: General Administration of Military Health, Tunisia (Network)
Responsible Party: Sponsor
Other Study IDs: UR17DN05SURVEY
Record Dates: First submitted 2021-02-04; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: HEALTH CARE WORKERS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to investigate the psychological impact of the COVID-19 outbreak on healthcare workers (HCWs) and to identify ways of coping with this unprecedented stressful situation.

DETAILED DESCRIPTION:
This was a cross-sectional study based on an online questionnaire that included 62 questions (scores, 0 - 3). The chi-square (χ²) test was used to compare the responses between professional groups, age groups, and genders.

ELIGIBILITY:
Inclusion Criteria:

* HEALTH CARE WORKERS

Exclusion Criteria:

* no one

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HEALTH CARE WORKERS all
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
STRESS-COVID | 01 months
  SURVEY ABOUT STRESS-COVID IN HEALTH CARE WORKERS

CONTACTS AND LOCATIONS:
Overall Officials: Hedi Gharsallah, MD, Study Chair — General Administration of Military Health, Tunisia
Locations (1):
- Military Hospital of Tunis, Tunis, Montfleury, Tunisia